CLINICAL TRIAL: NCT03461081
Title: An Open-label, Randomized, Two-sequence, Multiple-dose, Crossover Study to Evaluate Drug-drug Interaction Following Oral Administration of Telmisartan/Amlodipine and Atorvastatin in Healthy Adult Volunteers
Brief Title: Drug-drug Interaction Following Oral Administration of Telmisartan/Amlodipine and Atorvastatin in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JLP-1610-101-DDI
Record Dates: First submitted 2018-03-05; First posted 2018-03-09 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Hypertension With Hyperlipidemia
MeSH Terms: interventions — Telmisartan; Amlodipine; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Period I: administration of telmisartan/Amlodipine for 10 days then administration of telmisartan/amlodipine and atorvastatin for 4 days Period II: atorvastatin for 4 days
  Interventions: Drug: telmisartan/amlodipine and atorvastatin
- Group II (Experimental): Period I: administration of atorvastatin for 4 days Period II: administration of telmisartan/amlodipine for 10 days then administration of telmisartan/amlodipine and atorvastatin for 4 days
  Interventions: Drug: telmisartan/amlodipine and atorvastatin

INTERVENTIONS:
Drug: telmisartan/amlodipine and atorvastatin — Telmisartan/Amlodipine(40/5 mg) 2 Tab for 10 days Telmisartan/Amlodipine(40/5 mg) 2 Tab with Atorvastatin 40 mg 1 Tab for 4 days Atorvastatin 40 mg 1 Tab for 4 days

SUMMARY:
study to evaluate drug-drug interaction following oral administration of telmisartan/amlodipine and atorvastatin in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* 19~55 years healthy male
* The result of Body Mass Index(BMI) is not less than 19 kg/m2 , no more than 27 kg/m2
* Subjects who agree to keep contraceptive methods during the clinical trial.

Exclusion Criteria:

* Subjects who are allergic to investigational drug.
* Subjects who have a medical history which can affect the clinical trial.
* Hypertension(Systolic BP ≥ 150mmHG or Diastolic BP ≥ 100mmHg), Hypotension(Systolic BP ≤ 100mmHg or Diastolic BP ≤ 70mmHg)
* Liver enzyme (AST, ALT) level exceeds the maximum normal range more than one and a half times.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-07 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
AUCτ of telmisartan, amlodipine, atorvastatin, 2-OH atorvastatin | Period I Day 1, Day 10, Day 14 and Period II Day 4 pre and post 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24 hours
Css,max of telmisartan, amlodipine, atorvastatin, 2-OH atorvastatin | Period I Day 1, Day 10, Day 14 and Period II Day 4 pre and post 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No